CLINICAL TRIAL: NCT05050110
Title: Evaluation of Increased Fruits and Vegetables Consumption in Chronic Kidney Disease Patients Maintaining Normokalemia With Patiromer
Brief Title: Evaluation of Increased Fruits and Vegetables Consumption in Chronic Kidney Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nand Wadhwa (Other)
Responsible Party: Sponsor-Investigator, Nand Wadhwa, Nephrologist, Principal Investigator, NY Health d/b/a New York Cancer and Blood Specialists
Organization: NY Health d/b/a New York Cancer and Blood Specialists (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NYH-01
Record Dates: First submitted 2021-04-28; First posted 2021-09-20 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Fruit

STUDY DESIGN:
Intervention Model Description: Evaluation of Increased fruits and vegetables consumption in chronic kidney disease patients maintaining normokalemia with patiromer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic kidney disease patients (Other): Evaluation of Increased fruits and vegetables consumption in chronic kidney disease patients maintaining normokalemia with patiromer
  Interventions: Other: Fruits and Vegetable increase

INTERVENTIONS:
Other: Fruits and Vegetable increase — Increase fruits and vegetable consumption in chronic Kidney Patients to maintain Normokalemia

SUMMARY:
This study aims to investigate the feasibility of increasing dietary consumption of a rich variety of fruits and vegetables (including those that are potassim-rich) in patients with chronic kidney disease through use of nutritional counselling and hyperkalemia management with patiromer

DETAILED DESCRIPTION:
Adult Patients ages 18 and older with a diagnosis of Chronic Kidney Disease will be given a Diet Plan that consist of an increase of Fruits and Vegetables. Baseline data will be collected after the subject has signed the consent and their most recent eGFR and potassium level that is within 90 days has been reviewed to determine they are within the inclusion criteria.

Based on the approved Patiromer (Veltassa) package insert the subject will begin to take daily. During this control period of two weeks, the subject will document their normal daily consumption of fruits and vegetables in a provided food diary.

On the Second week, patient will receive dietary/nutritional counseling on the importance of potassium-rich fruits and vegetables. They will be instructed to increase their fruit and vegetable intake based on personal preferences and nutritional guides located inside the food diary. Choices will be documented daily in the supplied food diaries.

The Bowel Diary will be classified according to the Bristol Stool Chart and Quality of Life. Nutrition Survey Questionnaire will be documented in that supplied log.

At each subsequent visit, food diaries will be reviewed to evaluate fruit and vegetable consumption, vital signs will be documented and labs collected to measure effects on potassium metabolism. Bowel habits and questionnaires will be completed by the subject to determine how their diet has affected their quality of life.

Patiromer (Veltessa) dosing will be adjusted based on their serum potassium values following the approved drug brochure guidelines and at the discretion of the investigator.

Subject will return to the clinic at specified time points up to 52 weeks on study. The Patient can continue Veltassa while in the follow up period until week 52 at the discretion of the Principle Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years of age with chronic kidney disease and hyperkalemia
2. Chronic kidney disease is defined as eGFR 15-44ml/min/1.73m2
3. Documented hyperkalemia which is defined as serum potassium ≥ 5.0 mmol/L during the last 90 days
4. Diet evaluation for hyperkalemia (serum potassium ≥ 5.0) during the last 90 days
5. Patients receiving RASS inhibitors, beta-blockers, or diuretics to be on stable doses for 2 weeks
6. Patients already receiving patiromer are eligible

Exclusion Criteria:

1. Patients with a known allergy to patiromer
2. Patients currently taking other potassium controlling agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
By increasing the consumption of Fruits and Vegetable in their daily diet using the Nutritional Fruits and Vegetable Diary based off of the USDA Nutritive Value of foods and completing the Quality of Life Nutritional Questionnaire. | 3 years
  Participants will increase the Fruit and vegetable consumption by following a Diet plan listed in the Nutritional Diary provided to them by the study site in the beginning of the study while taking Patiromer (Veltassa). This will record their daily intake of 26-28 servings of fruit and vegetables weekly. The Nutritional diary lists a Diet Plan that measures the serving size of 26-28 servings of the fruits and vegetables. The measurement of fruits and vegetables has been calculated by the Nutritionist based off of the USDA Nutritive Value of foods and listed on the diary to explain the serving sizes and suggestions of meal plans.

SECONDARY OUTCOMES:
The Kidney Function levels will be tested at each visit from blood samples provided by the subject. | 3 years
  The Kidney Function blood test samples will be taken from the subject to show overall kidney health in Chronic Kidney Disease Patients by increasing their fruit and vegetable intake while on patiromer. The blood tests that support this is , Magnesium, phosphorus, iPTH, lipid panel, uric acid, hemoglobin A1C, Vitamin D 25(OH), Vitamin D 1,25(OH), FGF-23 and CBC panel.

OTHER OUTCOMES:
Measure the subjects diet intake related to Quality of Life | 3 years
  The subject will complete a Quality of Life Nutritional Questionnaire which is an instrument supported by ncbi to assess quality of life in relation to nutrition.
Measure the description of Daily bowel moments to test for constipation | 3 years
  Patient will complete a daily bowel Diary based on the Bristol Stool Chart which is a medical aid designed to classify feces into seven groups. The Diary will be provided to the subject to observe and classify their daily bowel movements.
Urine will be measured to evaluate kidney function in subjects with Chronic kidney disease | 3 years
  Tests will include 24 hour urine & Random for sodium, potassium, chloride, magnesium, phosphorus, calcium, urea nitrogen, creatinine, protein, albumin
Measure serum Potassium blood levels to remain below 5mmol/L | 3 years
  Serum Potassium levels are measured by blood samples from the subject that consists of either A Comprehensive Metabolic Panel blood test which includes or Basic Metabolic Panel depending on the timepoint in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nand Wadwha, MD, Principal Investigator — NY Health
Locations (1):
- NY Health, Port Jefferson Station, New York, United States